CLINICAL TRIAL: NCT05376917
Title: Quality of Life and Uncorrected Binocular Visual Acuity (UBVA) Evaluation in Patients Undergoing Cataract Surgery Using 4 Different Types of Lens Implant Combinations: a Multicenter, Prospective, Comparative and Randomized Study
Brief Title: Quality of Life Evaluation After Cataract Surgery Using 4 Types of Intraocular Lens Implant Combinations
Acronym: ELVIRA4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-03-CHRMT
Record Dates: First submitted 2022-03-28; First posted 2022-05-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cataract; Intraocular Lens Implant
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zeiss CT Asphina / Zeiss CT Asphina (Experimental): Monovision with refractive target of -1.50 Diopters (D) on the dominated eye
  Interventions: Device: Zeiss CT Asphina / Zeiss CT Asphina
- Zeiss AT Lara/ Zeiss AT Lisa Tri (Experimental): Zeiss AT Lara (dominant eye) / Zeiss AT Lisa Tri (non-dominant eye)
  Interventions: Device: Zeiss AT Lara/ Zeiss AT Lisa Tri
- Zeiss CT Asphina/ Zeiss AT Lara (Experimental): Zeiss CT Asphina/ Zeiss AT Lara (non-dominant eye)
  Interventions: Device: Zeiss CT Asphina/ Zeiss AT Lara
- Zeiss AT Lara / Zeiss AT Lara (Experimental): Micro-monovision with refractive target of -0.75 Diopters (D) on the non-dominant eye
  Interventions: Device: Zeiss AT Lara / Zeiss AT Lara

INTERVENTIONS:
Device: Zeiss CT Asphina / Zeiss CT Asphina — Monovision with refractive target of -1.50D on the dominated eye
  Arms: Zeiss CT Asphina / Zeiss CT Asphina
Device: Zeiss AT Lara/ Zeiss AT Lisa Tri — Zeiss AT Lara (dominant eye) / Zeiss AT Lisa Tri (non-dominant eye)
  Arms: Zeiss AT Lara/ Zeiss AT Lisa Tri
Device: Zeiss CT Asphina/ Zeiss AT Lara — Zeiss CT Asphina/ Zeiss AT Lara (non-dominant eye)
  Arms: Zeiss CT Asphina/ Zeiss AT Lara
Device: Zeiss AT Lara / Zeiss AT Lara — Micromonovision with refractive target of -0.75D on the non-dominant eye
  Arms: Zeiss AT Lara / Zeiss AT Lara

SUMMARY:
This is multicenter, prospective, comparative and randomized study focusing on the evolution of the quality of Life and Uncorrected Binocular Visual Acuity (UBVA) evaluation at 3 months after cataract surgery in patients who underwent 4 different types of intraocular lens Implant (IOL) combinations.

DETAILED DESCRIPTION:
Cataract, linked to the loss of transparency of the lens, is the leading cause of blindness in the world. It requires exclusively surgical treatment. Cataract surgery by ultrasonic phacoemulsification is the most common surgical procedure in France (800,000/year). The lens is removed and replaced with an artificial intraocular lens.

There are different types of implants that can be used. The simplest is the monofocal implant which is implanted in such a way as to correct "only far or near vision". For near vision or vice versa, it is therefore necessary to wear corrective lenses after the operation. A technique that eliminates the need for distance and near correction is based on monovision. This is a presbyopia compensation technique that aims to induce a slight myopization of one eye for near vision (usually the dominated eye) the other eye being intended for distance vision (dominant eye). There is therefore a difference in correction and perception of the images. Depending on the fixed distance, one eye will see sharp, the other less clear, even blurry. This difference can lead to a reduction in the perception of relief.

Other methods of compensating for presbyopia include the use of so-called multifocal or extended depth of field implants; they are also not devoid of sometimes annoying side effects (in particular possible halos around light sources at night) which can lead in rare cases to the removal of the intraocular lens.

However, patient requirements in terms of comfort of vision and independence from glasses are increasingly high and patients themselves are increasingly informed of the existence of multifocal implants. The choice of the intraocular implant to use is therefore a real challenge, especially since patients are often still active on a professional level.

Moreover, there is a lack of scientific consensus related to the choice of implants, during a surgical treatment of cataract lenses by phakoexeresis, for otherwise healthy eyes and in a subject wishing to no longer wear glasses postoperatively. . Different studies have emerged comparing the bilateral implantation of different types of multifocal implants with each other, but there is little work concerning mixed batches of "mix - match" implants.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from bilateral cataract and undergoing cataract surgery
* Patient with preoperative visual acuity ≤ 8/10th Monoyer (≥+ 0.1 logMar) in each eye
* Patient with nuclear color (NC), cortical (C) or posterior capsule opacity (P) cataract of normal to severe density in the Lens Opacities Classification System III (LOCSIII)
* Patient with cortical cataracts classified C1 to C5
* Patient with cataracts classified as nuclear opalescence (NO)1 to NO4 and nuclear color (NC)1 to NC4
* Patient with posterior capsule opacity cataracts classified as grade 5 (P1-P5)
* Patient affiliated to a social security scheme
* Patient having given written consent

Exclusion Criteria:

* Patient with biometrics ≤ 17 Diopters (D) and ≥ 28D
* Patient with a history (ATCD) of refractive surgery
* Patient with ATCD intraocular surgery
* Patient with ATCD strabismus
* Patient with amblyopia
* Patient with monophthalmos
* Patient with age-related macular degeneration (AMD)
* Patient with glaucoma
* Patient with diabetic retinopathy or maculopathy
* Patient with progressive or old ocular inflammatory disease
* Patient presenting with a very dense nuclear cataract (Stage NO5-6, NC5-6 on the LOCSIII classification), sources of preoperative complication
* Patient with keratoconus
* Patient with pseudoexfoliative syndrome
* Patient with pigment dispersion
* Patient with traumatic cataract
* Patient with astigmatism conforming to the rule > 1.5 Diopters (D) or inverse to the rule > 1 Diopter (D)
* Patient with abnormal ocular morphology
* Patient with abnormal keratometry
* Insulin-dependent diabetics and/or diabetics with retinal complications
* Pregnant or breastfeeding women
* Patient under legal protection (guardianship, curators, safeguard of justice)
* Person deprived of liberty
* Patient wishing to see near or far exclusively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
National Eye Institute Visual Functioning Questionnaire - 25 (NEI VFQ-25) questionnaire score before cataract surgery | Few days before surgery
  Quality of life score is obtained using the National Eye Institute Visual Functioning Questionnaire - 25 (NEI VQF-25) questionnaire score and measured before intervention.
  NEI VFQ-25 questionnaire measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases.
  The Visual Function Questionnaire (VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points (100 is the best score), respectively.
National Eye Institute Visual Functioning Questionnaire - 25 (NEI VFQ-25) questionnaire score 3 months after surgery | 3 months after surgery
  Quality of life score is obtained using the National Eye Institute Visual Functioning Questionnaire - 25 (NEI VQF-25) questionnaire score and measured 3 months after intervention.
  NEI VFQ-25 questionnaire measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases.
  The Visual Function Questionnaire-25 (VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points (100 is the best score), respectively.

SECONDARY OUTCOMES:
Uncorrected binocular visual acuity for far vision measured before intervention | Few days before surgery
  Uncorrected binocular visual acuity for distance vision is measured before intervention using Monoyer scale for far vision, scores ranging from 1 to 10, higher scores mean a better outcome; score 10 is the best.
Uncorrected binocular visual acuity for intermediate vision measured before intervention | Few days before surgery
  Uncorrected binocular visual acuity is measured before intervention using Parinaud scale for intermediate vision.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for near vision measured before intervention | Few days before surgery
  Uncorrected binocular visual acuity is measured before intervention using Parinaud scale for near vision.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for far vision measured 4 days postoperatively | 4 days after surgery
  Uncorrected binocular visual acuity for far vision is measured 4 days postoperatively using Monoyer scale for far vision, scores ranging from 1 to 10, higher scores mean a better outcome; score 10 is the best.
Uncorrected binocular visual acuity for intermediate vision measured 4 days postoperatively | 4 days after surgery
  Uncorrected binocular visual acuity for intermediate vision is measured 4 days postoperatively using Parinaud scale.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for far vision measured 1 month postoperatively | 1 month after surgery
  Uncorrected binocular visual acuity is measured 1 month after surgery using Monoyer scale for far vision, scores ranging from 1 to 10, higher scores mean a better outcome; score 10 is the best.
Uncorrected binocular visual acuity for intermediate vision measured 1 month postoperatively | 1 month after surgery
  Uncorrected binocular visual acuity is measured 1 month after surgery using Parinaud scale.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for near vision measured 1 month postoperatively | 1 month after surgery
  Uncorrected binocular visual acuity is measured 1 month after surgery using Parinaud scale.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for far vision measured 3 months postoperatively | 3 months after surgery
  Uncorrected binocular visual acuity is measured 3 months after surgery using Monoyer scale for far vision, scores ranging from 1 to 10, higher scores mean a better outcome; score 10 is the best.
Uncorrected binocular visual acuity for intermediate vision measured 3 months postoperatively | 3 months after surgery
  Uncorrected binocular visual acuity for intermediate vision is measured 3 months after surgery using Parinaud scale.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Uncorrected binocular visual acuity for near vision measured 3 months postoperatively | 3 months after surgery
  Uncorrected binocular visual acuity for near vision is measured 3 months after surgery using Parinaud scale.
  The Parinaud scale ranges from Parinaud 14 (P 14) (lowest score) to Parinaud 1.5 (P 1.5) (best score).
Sunglasses wear frequency 3 months after surgery for far and near visions | 3 months after surgery
  Frequency of wearing sunglasses in patients undergoing IOL implant surgery : permanently (yes/no) or occasionally (yes/no) for far and near visions
Eye tonicity before surgery | Few days before surgery
  Eye pressure measurement millimeters of mercury (mmHg) before intervention
Eye tonicity 4 days postoperatively | 4 days after surgery
  Eye pressure measurement millimeters of mercury (mmHg) 4 days postoperatively
Eye tonicity 1 month postoperatively | 1 month after surgery
  Eye pressure measurement millimeters of mercury (mmHg) 1 month postoperatively
Eye tonicity 3 months postoperatively | 3 months after surgery
  Eye pressure measurement millimeters of mercury (mmHg) 3 months postoperatively
Slit lamp and Macular Optical coherence tomography (OCT) examination before surgery | Few days before surgery
  Presence of postoperative complications: Persistent lens mass (Yes/No); Tyndall effect (Yes/No) Hyphema (Yes/No); Irian hernia (Yes/No); Endophthalmitis (Yes/No); Implant dislocation (Yes/No)
Slit lamp and Macular OCT examination 4 days postoperatively | 4 days after surgery
  Presence of postoperative complications: Persistent lens mass (Yes/No); Tyndall effect (Yes/No) Hyphema (Yes/No); Irian hernia (Yes/No); Endophthalmitis (Yes/No); Implant dislocation (Yes/No)
Slit lamp and Macular OCT examination 1 month postoperatively | 1 month after surgery
  Presence of postoperative complications: Persistent lens mass (Yes/No); Tyndall effect (Yes/No); Hyphema (Yes/No); Irian hernia (Yes/No); Endophthalmitis (Yes/No); Implant dislocation (Yes/No)
Slit lamp and Macular OCT examination 3 months postoperatively | 3 months after surgery
  Presence of postoperative complications: Persistent lens mass (Yes/No); Tyndall effect (Yes/No); Hyphema (Yes/No); Irian hernia (Yes/No); Endophthalmitis (Yes/No); Implant dislocation (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc PERONE, MD, Principal Investigator — Mercy Hospital CHR Metz Thionville
Locations (2):
- France (2):
  - CHR Metz-Thionville/Hopital de Mercy, Metz
  - CHR Metz-Thionville_Hopital Bel Air, Metz